CLINICAL TRIAL: NCT03929744
Title: A Single- and Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3502970 in Healthy Subjects
Brief Title: A Study of LY3502970 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 17416; J2A-MC-GZGA (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-04-25; First posted 2019-04-29 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Healthy
MeSH Terms: interventions — orforglipron; Atorvastatin; Simvastatin; Midazolam

STUDY DESIGN:
Intervention Model Description: Part C is a crossover design.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- LY3502970 (Part A) (Experimental): Single dose of LY3502970 administered orally.
  Interventions: Drug: LY3502970
- Placebo (Part A) (Placebo Comparator): Single dose of placebo administered orally.
  Interventions: Drug: Placebo
- LY3502970 (Part B) (Experimental): Multiple doses of LY3502970 administered orally. Some participants will also receive atorvastatin and simvastatin or midazolam administered orally.
  Interventions: Drug: LY3502970; Drug: Atorvastatin; Drug: Simvastatin; Drug: Midazolam
- Placebo (Part B) (Placebo Comparator): Multiple doses of placebo administered orally. Some participants will also receive atorvastatin and simvastatin or midazolam administered orally.
  Interventions: Drug: Placebo; Drug: Atorvastatin; Drug: Simvastatin; Drug: Midazolam
- LY3502970 (Part C) (Experimental): Single dose of LY3502970 administered orally in each of two study periods.
  Interventions: Drug: LY3502970
- LY3502970 (Part D) (Experimental): Single dose of LY3502970 administered orally.
  Interventions: Drug: LY3502970
- Placebo (Part D) (Placebo Comparator): Single dose of placebo administered orally.
  Interventions: Drug: Placebo
- LY3502970 Formulation 1 (Part E) (Experimental): Multiple doses of LY3502970 - formulation 1 administered orally.
  Interventions: Drug: LY3502970
- LY3502970 Formulation 2 (Part E) (Experimental): Multiple doses of LY3502970 - formulation 2 administered orally.
  Interventions: Drug: LY3502970

INTERVENTIONS:
Drug: LY3502970 — Administered orally.
  Arms: LY3502970 (Part A); LY3502970 (Part B); LY3502970 (Part C); LY3502970 (Part D); LY3502970 Formulation 1 (Part E); LY3502970 Formulation 2 (Part E)
Drug: Placebo — Administered orally.
  Arms: Placebo (Part A); Placebo (Part B); Placebo (Part D)
Drug: Atorvastatin — Administered orally.
  Arms: LY3502970 (Part B); Placebo (Part B)
Drug: Simvastatin — Administered orally.
  Arms: LY3502970 (Part B); Placebo (Part B)
Drug: Midazolam — Administered orally.
  Arms: LY3502970 (Part B); Placebo (Part B)

SUMMARY:
The main purposes of this study are to determine:

* The safety of LY3502970 and any side effects that might be associated with it.
* How much LY3502970 gets into the bloodstream and how long it takes the body to get rid of it.

This study has 5 parts (A, B, C, D, and E). Parts A and D involve a single dose of LY3502970 and will last about 15 days. Part B and E involve multiple doses of LY3502970 and will last about 4 weeks. Part C involves two single doses of LY3502970 and will last about 29 days. Each participant will enroll in only one part. Screening must be completed within 28 days before study start. This study is for research purposes only, and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females, as determined by medical history
* Have safety laboratory results within normal reference ranges

Exclusion Criteria:

* Have known allergies to LY3502970, glucagon-like peptide-1 (GLP-1) analogs, related compounds
* Abnormal electrocardiogram (ECG) at screening
* Significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological or neurological disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug | Baseline up to Day 42
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3502970 | Predose up to 96 hours postdose
  PK: Cmax of LY3502970
PK: Area Under the Concentration Versus Time Curve from Time Zero to the Last Measurable Concentration (AUC[0-tlast]) of LY3502970 | Predose up to 96 hours postdose
  PK: AUC(0-tlast) of LY3502970
PK: Time of Maximum Observed Concentration (Tmax) of LY3502970 | Predose up to 96 hours postdose
  PK: Tmax of LY3502970

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma X, Liu R, Pratt EJ, Benson CT, Bhattachar SN, Sloop KW. Effect of Food Consumption on the Pharmacokinetics, Safety, and Tolerability of Once-Daily Orally Administered Orforglipron (LY3502970), a Non-peptide GLP-1 Receptor Agonist. Diabetes Ther. 2024 Apr;15(4):819-832. doi: 10.1007/s13300-024-01554-1. Epub 2024 Feb 24. PMID 38402332